CLINICAL TRIAL: NCT06962670
Title: Digital and Molecular Detection of Markers for Disease Risk Prediction, Improvement of Diagnostic Detection Accuracy and Implementation for Preventive Measures of Cancer - A Combined Case-control and Cohort Study
Brief Title: Predicting Cancer Risk With Digital and Molecular Markers
Acronym: PräDigt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Peter A. Fasching, Prof. Dr. med., University Hospital Erlangen
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PräDigt-08/22
Record Dates: First submitted 2023-08-23; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case group (subjects with known pre-existing or current cancer diagnosis) (Other): The case group will consist of subjects with a known pre-existing or current cancer diagnosis, including breast cancer, lung cancer, colorectal cancer or gynecologic cancer
  Interventions: Other: Biomaterial collection; Other: BayPass mobile application
- Control group (healthy subjects) (Other): The control group will consist of healthy subjects with no history of cancer
  Interventions: Other: Biomaterial collection; Other: BayPass mobile application

INTERVENTIONS:
Other: Biomaterial collection — All subjects will be asked to provide biomaterial (blood or saliva) for bio marker screening and analysis. Additional biomaterial (breath, urin, stool) is optional.
Other: BayPass mobile application — All subjects will be asked to use the study-specific mobile application "BayPass" to complete questionnaires and provide results from screening examinations over a course of 12 months.

SUMMARY:
The goal of this study is to identify new markers to predict the risk of developing cancer, primarily breast cancer. For this purpose, researchers will compare data obtained from cancer patients and healthy individuals. If characteristic differences are identified, e.g. in biomarkers, life style or family history, this may indicate a person's increased risk of developing cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Biological adult (at least 18 years old) women
2. Written informed consent for study participation and processing of personal data
3. Own smartphone that can run the BayPass mobile application and willingness to use said smartphone for study purposes

   Additional inclusion criterion for case group:
4. Pre-existing or current diagnosis of at least one of the following oncological diseases: breast cancer, lung cancer, colorectal cancer, gynecologic cancer (incl. ovarian cancer, endometrial cancer, cervical cancer, fallopian tube cancer, vaginal cancer and vulvar cancer)

Exclusion Criteria:

1. Known infection with HIV (Human Immunodeficiency Virus), HepA (Hepatitis A), HepB (Hepatitis B), HepC (Hepatitis C) or active SARS-CoV2 (Severe acute respiratory syndrome coronavirus type 2) infection
2. Acute severe or potentially life-threatening illness, except those specified in inclusion criterion #4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of breast cancer risk by polygenic risk score in combination with app-based self-reported health behavior in the study population | Baseline
  Polygenic cancer risk score (PRS) as a numeric value using BOADICEA/CanRisk as absolute 10-year breast cancer risk and as relative risk compared with avarage women at the same age

CONTACTS AND LOCATIONS:
Overall Officials: Matthias W. Beckmann, Prof. Dr. med., Study Director — Head of Department of Obstetrics and Gynecology
Locations (1):
- DigiOnko Präventionsmobil, Please Refer to Project Homepage For Details (see Link Below), Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: On this project homepage you can check where the next stop of the DigiOnko Präventionsmobil will be — https://www.digionko-bayern.de/praeventionsmobil/